CLINICAL TRIAL: NCT05352165
Title: A Prospective Multicenter Randomized Controlled Trial of the Clinical Efficacy of Neoadjuvant Therapy Based on Organoids Drug Sensitivity Versus Empirical Neoadjuvant Therapy in the Treatment of Advanced Rectal Cancer
Brief Title: The Clinical Efficacy of Drug Sensitive Neoadjuvant Chemotherapy Based on Organoid Versus Traditional Neoadjuvant Chemotherapy in Advanced Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Collaborators: Shanghai OneTar Biomedicine Co., Ltd. (Unknown); Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MISC-WXXR-001
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Neoadjuvant Therapy
Keywords: neoadjuvant therapy; organoid drug sensitivity; advanced rectal cancer
MeSH Terms: interventions — Folfox protocol; Fluorouracil; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is a prospective multicenter multi-arm umbrella clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- standard long-term therapy (Experimental): The standard whole-course neoadjuvant therapy group was treated with neoadjuvant simultaneous radiotherapy and chemotherapy (Total Neoadjuvant Therapy, TNT) based on guidelines and clinical experience.
  Interventions: Drug: standard long-term therapy; Drug: FOLFOX and standard long-term radiotherapy; Drug: FOLFIRI and standard long-term radiotherapy; Drug: 5-FU and standard long-term radiotherapy; Drug: 5-FU and pembrolizumab and standard long-term radiotherapy; Drug: Other individualized treatments
- FOLFOX and standard long-term radiotherapy (Active Comparator): FOLFOX and standard long-term radiotherapy based on organoids drug sensitivity
  Interventions: Drug: standard long-term therapy; Drug: FOLFOX and standard long-term radiotherapy; Drug: FOLFIRI and standard long-term radiotherapy; Drug: 5-FU and standard long-term radiotherapy; Drug: 5-FU and pembrolizumab and standard long-term radiotherapy; Drug: Other individualized treatments
- FOLFIRI and standard long-term radiotherapy (Active Comparator): FOLFIRI and standard long-term radiotherapy based on organoids drug sensitivity
  Interventions: Drug: standard long-term therapy; Drug: FOLFOX and standard long-term radiotherapy; Drug: FOLFIRI and standard long-term radiotherapy; Drug: 5-FU and standard long-term radiotherapy; Drug: 5-FU and pembrolizumab and standard long-term radiotherapy; Drug: Other individualized treatments
- 5-FU and standard long-term radiotherapy (Active Comparator): 5-FU and standard long-term radiotherapy based on organoids drug sensitivity
  Interventions: Drug: standard long-term therapy; Drug: FOLFOX and standard long-term radiotherapy; Drug: FOLFIRI and standard long-term radiotherapy; Drug: 5-FU and standard long-term radiotherapy; Drug: 5-FU and pembrolizumab and standard long-term radiotherapy; Drug: Other individualized treatments
- 5-FU and pembrolizumab and standard long-term radiotherapy (Active Comparator): 5-FU and pembrolizumab and standard long-term radiotherapy based on organoids drug sensitivity
  Interventions: Drug: standard long-term therapy; Drug: FOLFOX and standard long-term radiotherapy; Drug: FOLFIRI and standard long-term radiotherapy; Drug: 5-FU and standard long-term radiotherapy; Drug: 5-FU and pembrolizumab and standard long-term radiotherapy; Drug: Other individualized treatments
- Other individualized treatments (Active Comparator): Other individualized treatments based on organoids drug sensitivity
  Interventions: Drug: standard long-term therapy; Drug: FOLFOX and standard long-term radiotherapy; Drug: FOLFIRI and standard long-term radiotherapy; Drug: 5-FU and standard long-term radiotherapy; Drug: 5-FU and pembrolizumab and standard long-term radiotherapy; Drug: Other individualized treatments

INTERVENTIONS:
Drug: standard long-term therapy — The standard whole-course neoadjuvant therapy group was treated with neoadjuvant simultaneous radiotherapy and chemotherapy (Total Neoadjuvant Therapy, TNT) based on guidelines and clinical experience.
Drug: FOLFOX and standard long-term radiotherapy — FOLFOX and standard long-term radiotherapy based on organoids drug sensitivity
Drug: FOLFIRI and standard long-term radiotherapy — FOLFIRI and standard long-term radiotherapy based on organoids drug sensitivity
Drug: 5-FU and standard long-term radiotherapy — 5-FU and standard long-term radiotherapy based on organoids drug sensitivity
Drug: 5-FU and pembrolizumab and standard long-term radiotherapy — 5-FU and pembrolizumab and standard long-term radiotherapy based on organoids drug sensitivity
Drug: Other individualized treatments — Other individualized treatments based on organoids drug sensitivity

SUMMARY:
This is a prospective multicenter randomized controlled trial study. According to the enrollment criteria, patients with locally advanced rectal cancer who need neoadjuvant therapy before radical surgery were randomly divided into the organoids drug sensitivity group and the standard whole-course neoadjuvant therapy group. The Organoids drug sensitivity group was treated with personalized neoadjuvant therapy under the guidance of tumor organoids drug sensitivity technology combined with standard long-term radiotherapy. The standard whole-course neoadjuvant therapy group was treated with neoadjuvant simultaneous radiotherapy and chemotherapy (Total Neoadjuvant Therapy, TNT) based on guidelines and clinical experience. The tumor pathological complete remission rate (pCR), postoperative complication rate, postoperative tumor withdrawal grade, postoperative recurrence rate, treatment tolerance rate, R0 resection rate, and sphincter preservation rate were observed and compared.

DETAILED DESCRIPTION:
Based on the need for individualized treatment in the era of precision medicine, an in vitro model that can accurately predict the response of patients to treatment is urgently needed, so that suitable patients can receive effective treatment and patients whose treatments are ineffective can avoid adverse reactions. The emergence of tumor organoids technology makes this vision possible.

Tumor-organoid (Patient-Derived Organoids, PDOs) is a kind of micro-organ with a three-dimensional structure, which is cultivated in the environment of 3D matrix glue in vitro. Based on the individualized neoadjuvant therapy based on the drug sensitivity technology of tumor-organoid, the best neoadjuvant therapy can be selected and the clinical efficacy and drug tolerance can be quickly predicted, which is of great significance in the field of accurate tumor therapy. The preliminary study of our group also completed the organ-like library of more than 100 patients with local advanced rectal cancer. It was proved that the organoids of the organoids library had high homology with the original tumor tissue, and the detection period of drug sensitivity of organoids was less than 2 weeks, which was much less than 2 months of PDX drug sensitivity technology in mice, which did not affect the time window of clinical drug treatment, and the results of drug sensitivity were basically consistent with the clinical efficacy.

Therefore, we have reason to believe that tumor organoids chemosensitivity technology, as an economical, high-throughput, and efficient technology for tumor research, is expected to play an important role in clinical individualized treatment of tumors.

Our previous study found that tumor-based organoids drug sensitivity technology can be used as an effective and reliable clinical assistant tool to guide and assist doctors to formulate the best treatment strategy for tumor patients. Personalized neoadjuvant therapy has better clinical efficacy than standard whole-course neoadjuvant therapy.

Therefore, in this study, through a prospective, multicenter, multi-arm umbrella clinical study, patients with locally advanced rectal cancer who need neoadjuvant therapy are randomly divided into two groups: the organoids drug sensitivity group and the standard whole-course neoadjuvant therapy group. To compare the clinical efficacy of personalized neoadjuvant therapy based on tumor organoids chemosensitivity combined with standard long-term radiotherapy with the clinical efficacy of standard whole-course neoadjuvant therapy in locally advanced rectal cancer. This technology can be used in the clinical use of advanced rectal cancer new auxiliary decision-making system so that the standardization of comprehensive treatment of rectal cancer can be implemented in China, which is of great significance for the development of the national economy and the improvement of medical level in China.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age: 18-75. 2) qualitative diagnosis: adenocarcinoma was confirmed by enteroscopic biopsy. 3) Localization diagnosis: the tumor is located in the rectum (the distance between the tumor and the anal margin ≤ 12cm).

  4) plain scan of thoracoabdominal pelvis and enhanced CT or MRI evaluation of rectal cancer staging:

The primary tumor invades the muscular layer of the intestinal wall into the surrounding well-known structure, with or without lymph node metastasis in the proper rectal fascia.

b. TNM clinical or pathological stage of tumor: T3-T4N0-2M0. 5) physical condition (ECOG) score ≤ 1. 6) all patients agreed to receive adjuvant chemotherapy for 3 to 6 months after operation.

7) sign informed consent and participate in the project voluntarily.

Exclusion Criteria:

* 1) simultaneous or metachronous multiple primary malignant tumors. 2) preoperative imaging examination or pathological results showed that:

Lateral lymph node metastasis. b. Distant organ metastasis. 3) previous history of malignant tumors. 4) abnormal function of heart, lung, liver, kidney, hematopoiesis and bone marrow reserve, which can not tolerate neoadjuvant therapy and operation.

5) have mental illness or other serious cardiovascular disease. 6) pregnant or lactating women. 7) Emergency surgery (perforation, bleeding, intestinal obstruction, etc.). 8) BRAF mutation was found by gene detection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response | 3 years
  Neoadjuvant therapy and postoperative pathology confirmed that the primary tumor was in complete remission (stage ypT0) and had no residual tumor cells, regardless of whether the regional lymph nodes were involved or not.

SECONDARY OUTCOMES:
Postoperative complication | 3 years
  Intra-abdominal bleeding, anastomotic leakage, intra-abdominal infection, intestinal obstruction, postoperative diarrhea, wound infection, pulmonary infection, cardiovascular accident, cerebrovascular accident, etc.
Tumor Regression Grading | 3 years
  Tumor pathological reaction is graded after neoadjuvant therapy, usually according to the proportion of fibrosis and residual tumor in the tumor.
  The analytical system for evaluating treatment response recommended by NCCN is as follows: complete response-no living cancer cell residue, moderate reaction-single or small cluster cancer cell residue,mild reaction-residual cancer focus, interstitial fibrosi,adverse reaction-few or no cancer cell regression.
Local recurrence | 3 years
  Recurrence occurs in the surgical area, with or without the rise of tumor markers. The tumor found in the anastomosis needs to be confirmed by pathological biopsy.
Distant metastasis | 3 years
  CT or MRI or radionuclide scan can detect metastases in liver, lung and bone, with or without confirmed by pathology.
Treatment tolerance rate | 3 years
  To evaluate the tolerance and completion of preoperative neoadjuvant therapy.
R0 resection rate | 3 years
  R0 resection rate of laparoscopic radical surgery for rectal cancer after neoadjuvant therapy.
anus-saving rate | 3 years
  anus-saving rate after radical resection of rectal cancer after neoadjuvant therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jing Sun, PhD, Principal Investigator — Shanghai Minimally Invasive Surgery Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA Cancer J Clin. 2021 Jan;71(1):7-33. doi: 10.3322/caac.21654. Epub 2021 Jan 12. PMID 33433946
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Cao W, Chen HD, Yu YW, Li N, Chen WQ. Changing profiles of cancer burden worldwide and in China: a secondary analysis of the global cancer statistics 2020. Chin Med J (Engl). 2021 Mar 17;134(7):783-791. doi: 10.1097/CM9.0000000000001474. PMID 33734139
- [Background] Ludmir EB, Palta M, Willett CG, Czito BG. Total neoadjuvant therapy for rectal cancer: An emerging option. Cancer. 2017 May 1;123(9):1497-1506. doi: 10.1002/cncr.30600. Epub 2017 Mar 10. PMID 28295220
- [Background] Garcia-Aguilar J, Chow OS, Smith DD, Marcet JE, Cataldo PA, Varma MG, Kumar AS, Oommen S, Coutsoftides T, Hunt SR, Stamos MJ, Ternent CA, Herzig DO, Fichera A, Polite BN, Dietz DW, Patil S, Avila K; Timing of Rectal Cancer Response to Chemoradiation Consortium. Effect of adding mFOLFOX6 after neoadjuvant chemoradiation in locally advanced rectal cancer: a multicentre, phase 2 trial. Lancet Oncol. 2015 Aug;16(8):957-66. doi: 10.1016/S1470-2045(15)00004-2. Epub 2015 Jul 14. PMID 26187751
- [Background] Shamir ER, Ewald AJ. Three-dimensional organotypic culture: experimental models of mammalian biology and disease. Nat Rev Mol Cell Biol. 2014 Oct;15(10):647-64. doi: 10.1038/nrm3873. Epub 2014 Sep 17. PMID 25237826
- [Background] Sato T, Vries RG, Snippert HJ, van de Wetering M, Barker N, Stange DE, van Es JH, Abo A, Kujala P, Peters PJ, Clevers H. Single Lgr5 stem cells build crypt-villus structures in vitro without a mesenchymal niche. Nature. 2009 May 14;459(7244):262-5. doi: 10.1038/nature07935. Epub 2009 Mar 29. PMID 19329995